CLINICAL TRIAL: NCT02504528
Title: Bronchial Provocation Tests With House Dust Mite in Allergic Asthma in Guangzhou
Brief Title: Bronchial Allergen Provocation Tests in Asthmatics in Guangzhou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Firestone Institute for Respiratory Health (Other)
Responsible Party: Principal Investigator, Jinping Zheng, Deputy director,GRID, Guangzhou Institute of Respiratory Disease
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GIRD201534; BAPT201534 (Registry Identifier: BAPT201534)
Record Dates: First submitted 2015-07-08; First posted 2015-07-22 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Allergic Asthma
Keywords: asthma; allergy; bronchial hyperresponsiveness; provocation
MeSH Terms: conditions — Asthma; Hypersensitivity; Bronchial Hyperreactivity | interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- allergic asthma (Experimental): asthma patients that sensitive to house dust mites.
  Interventions: Other: house dust mites
- normal controls (Experimental): normal controls with or without sensitive to house dust mites.
  Interventions: Other: house dust mites

INTERVENTIONS:
Other: house dust mites — house dust mites(two-fold increasing concentration of house dust mite (HDM) extract, dilutions prepared starting from 1:8, 1:16, 1:32, 1:64, 1:128, 1: 256, 1:512, 1:1024,……)

SUMMARY:
The purpose of this study is to establish the methodology of bronchial provocation tests with house dust mites in China, and to evaluate its safety and effects on upper and lower airways inflammation.

DETAILED DESCRIPTION:
After screening,each participant undergo baseline lung function test,airway inflammation evaluation (blood and sputum eosinophils count,interleukin-13 (IL-13),FeNO)and airway responsiveness tests(methacholine bronchial provocation,nasal histamine provocation).

On the second day,the participant undergo bronchial house dust mites challenge tests.

On the third day,the participant undergo the lung function test,airway inflammation evaluation (blood and sputum eosinophils count,IL-13,FeNO)and airway responsiveness tests(methacholine bronchial provocation,nasal histamine provocation).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma;
* Sensitive to house dust mite;
* Stable for more than 4 weeks with FEV1≥70%pred

Exclusion Criteria:

* exacerbation within 3 months;
* upper airway infections within 6 weeks;
* concomitant of hypertension or heart diseases;
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-01; Primary Completion 2017-07-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
percentages of the participants that tested positive to house dust mites bronchial provocation | 30 minutes after house dust mites bronchial provocation

SECONDARY OUTCOMES:
Changes of the percentages of eosinophils in sputum, nasal lavage and fractional exhaled nitric oxide (FeNO) from baseline | 30mins, 7 and 24 hours after bronchial challenge
Changes of provocative concentration induced a 20% decrease in forced expiratory volume at one second (FEV1) to methacholine before and after house dust mites bronchial provocation | 24 hours after house dust mites bronchial challenge
percentages of the participants that tested positive to house dust mites bronchial provocation measured by impulse oscillometry | 10 minutes after house dust mites bronchial provocation
Changes of provocative concentration induced a 60% increase in nasal airway resistance to histamine before and after house dust mites bronchial provocation | 24 hours after house dust mites bronchial challenge
  By Comparison with methacholine provocation test

OTHER OUTCOMES:
correlate of IL-4,IL-13,periostin with provocative concentration induced a 20% decrease in FEV1 to house dust mite in asthmatic | 30 mins and 24 hours after house dust mites bronchial challenge
  By Comparison with methacholine provocation test
Incidence and Severity of Adverse Events During The House Dust Mite Bronchial Provocation Test | 30 minutes, 7 hours and 24 hours after house dust mites bronchial provocation
  By Comparison with methacholine provocation test at 30 min and 24 hours after challenge test.

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, Principal Investigator — State Key Laboratory of Respiratory Disease; China Clinical Research Center of Respiratory Disease; First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China